CLINICAL TRIAL: NCT02093442
Title: Endometrial Scratching for Cryopreserved Embryo Transfer: a Randomized Controlled Trial
Brief Title: Endometrial Scratching for Cryopreserved Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The main investigators are no longer working at the center.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Wellington P Martins, MD, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAAE:03292412.0.0000.5440
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial injury (Experimental): Women allocated to this group will be submitted to endometrial injury before undergoing endometrial preparation for embryo transfer.
  Interventions: Procedure: Endometrial injury
- Control (No Intervention): Women allocated to this group will NOT be submitted to endometrial injury before undergoing endometrial preparation for embryo transfer.

INTERVENTIONS:
Procedure: Endometrial injury — Endometrial biopsy using a pipelle de Cornier
  Other Names: Endometrial scratching
  Arms: Endometrial injury

SUMMARY:
Endometrial injury performed in a cycle preceding the one for embryo transfer is associated with an increased implantation and pregnancy rate when carried out during the month preceding that of ovulation induction and fresh embryo transfer. However, there is no evidence about the effect of this intervention on the transfer of cryopreserved embryos.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* At least one cryopreserved embryo

Exclusion Criteria:

* None

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Live birth | 10 months
  The complete expulsion or extraction from its mother of a product of fertilization, irrespective of the duration of the pregnancy, which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation, or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.

SECONDARY OUTCOMES:
Clinical pregnancy | 3 months
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy. Note: Multiple gestational sacs are counted as one clinical pregnancy.
Miscarriage | 5 months
  The spontaneous loss of a clinical pregnancy

OTHER OUTCOMES:
Multiple pregnancy | 3 months
  A pregnancy with more than one gestational sac.

CONTACTS AND LOCATIONS:
Overall Officials: Wellington P Martins, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Setor de Reprodução Humana - FMRP-USP, Ribeirão Preto, São Paulo, Brazil